CLINICAL TRIAL: NCT00406055
Title: Carotid Stenting For High Surgical-Risk Patients; Evaluating Outcomes Through The Collection Of Clinical Evidence
Brief Title: CHOICE: Carotid Stenting For High Surgical-Risk Patients
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-717
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Provide an ongoing post-market surveillance mechanism for documentation of clinical outcomes and for possible extension of the Centers for Medicare and Medicaid Services (CMS) coverage to a broader group of patients.
  Interventions: Device: RX ACCULINK , RX ACCUNET , XACT , EMBOSHIELD and EMBOSHIELD Nav6

INTERVENTIONS:
Device: RX ACCULINK , RX ACCUNET , XACT , EMBOSHIELD and EMBOSHIELD Nav6 — Provide an ongoing post-market surveillance mechanism for documentation of clinical outcomes and for possible extension of the Centers for Medicare and Medicaid Services (CMS) coverage to a broader group of patients.

SUMMARY:
The purposes of this study is to 1) Provide additional information that the commercially available Abbott Vascular Carotid Stent Systems and Embolic Protection Systems can be used successfully by a wide range of physicians under commercial use conditions. 2) Provide an ongoing post-market surveillance mechanism for documentation of clinical outcomes and for possible extension of the Centers for Medicare and Medicaid Services (CMS) coverage to a broader group of patients.

DETAILED DESCRIPTION:
The CHOICE study will provide a mechanism for collection of data from Abbott Vascular's Carotid Stent Systems and Embolic Protection Systems when used by a broad group of physicians under commercial use conditions. The original CAPTURE and EXACT studies had built-in features that limited the ability to collect on-going real world data because they restricted the number of sites that could participate (up to 150 sites) and limited enrollment at each site (up to 50 patients per site). This study will not have these restrictions. The CHOICE study will also provide an ongoing post-market surveillance mechanism for documentation of clinical outcomes and for possible extension of the Centers for Medicare and Medicaid Services (CMS) coverage to a broader group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or patient's legally authorized representative provided informed consent.
2. Patient is considered at high risk for carotid endarterectomy (CEA).
3. Patient requires percutaneous carotid angioplasty and stenting for carotid artery disease.
4. Patients physician intends to use an RX Acculink with either the RX Accunet or Emboshield Nav 6 in the carotid artery OR the patients physician intends to use an Xact with the Emboshield or Emboshield Nav6 in the carotid artery as per the FDA approved Indications for Use as outlined.

Exclusion Criteria:

There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled into this registry will be male and female patients derived from the general population who satisfy the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 18855 (Actual)
Dates: Start 2006-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Composite of death, stroke, and MI (DSMI) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, M.D., Study Chair
Locations (1):
- Abbott Vascular, Santa Clara, California, United States